CLINICAL TRIAL: NCT04707118
Title: Peritoneal Perfusion Chemotherapy Combined With Gemcitabine and Albumin Binding Paclitaxel Versus Gemcitabine and Albumin Binding Paclitaxel in the Treatment of Advanced Pancreatic Cancer With Intraperitoneal Metastasis
Brief Title: Ntraperitoneal Thermal Perfusion Combined With Chemotherapy Versus Chemotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, President of Shanghai Pancreatic Cancer Institute, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-30
Record Dates: First submitted 2021-01-10; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Advanced Pancreatic Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal perfusion cisplatin+Nab-paclitaxel+GEM (Experimental): Laparoscopic exploration + thermal perfusion cisplatin 40 mg/m2, Postoperative exploration D1, 8 Nab-paclitaxel 125 mg/m2, GEM 1000 mg/m2, D1, 8, 15 after the second thermal perfusion 4 weeks plan, 6 cycles
  Interventions: Drug: cisplatin+Nab-paclitaxel+GEM
- Nab-paclitaxel+GEM (Active Comparator): Nab-paclitaxel 125 mg/m2, GEM 1000 mg/m2, D1, 8, 15 4 weeks plan, 6 cycles
  Interventions: Drug: Nab-paclitaxel+GEM

INTERVENTIONS:
Drug: cisplatin+Nab-paclitaxel+GEM — Laparoscopic exploration + thermal perfusion cisplatin 40 mg/m2, Postoperative exploration D1, 8 Nab-paclitaxel 125 mg/m2, GEM 1000 mg/m2, D1, 8, 15 after the second thermal perfusion 4 weeks plan, 6 cycles
  Arms: Thermal perfusion cisplatin+Nab-paclitaxel+GEM
Drug: Nab-paclitaxel+GEM — Nab-paclitaxel 125 mg/m2, GEM 1000 mg/m2, D1, 8, 15 4 weeks plan, 6 cycles
  Arms: Nab-paclitaxel+GEM

SUMMARY:
In view of the existence of malignant ascites in patients with advanced pancreatic cancer, we put forward the heat abdominal cavity perfusion chemotherapy combined albumin paclitaxel and gemcitabine compared with albumin paclitaxel and gemcitabine prospective clinical study, to assess abdominal albumin hot perfusion chemotherapy combined control of ascites and taxol in improving patients' quality of life, survival, exploring the feasibility of celiac hot perfusion chemotherapy combined albumin paclitaxel and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participate voluntarily and sign informed consent;
* Age ≥18 years old and ≤80 years old, regardless of gender;
* Physical condition ECOG 0 ~ 2;
* The diagnosis of pancreatic adenocarcinoma was confirmed by pathology;
* Peritoneal metastasis was confirmed by ascites cytology, or was pathologically confirmed by surgical exploration and biopsy;
* Expected survival ≥3 months;
* No serious abnormal blood system, heart and lung function and immune deficiency (refer to respective standards);
* Blood routine indicators: white blood cell (WBC) ≥3 × 109/L;Absolute count of neutrophils (ANC) ≥1.5 × 109/L;Platelet (PLT) ≥100 × 109/L;Hemoglobin (Hgb) ≥9 g/dL;
* Blood biochemical indexes: AST (SGOT) and ALT (SGPT) ≤2.5 × upper limit of normal value (ULN);Total bilirubin (TBIL) ≤ULN;Serum creatinine (CRE) ≤1.5 × ULN;
* Coagulation function: Prothrombin time (PT), international standard ratio (INR) ≤1.5 × ULN;
* Comply with the study visit plan and other program requirements.

Exclusion Criteria:

* Accompanied by other systemic malignant tumors;
* Received any form of anti-tumor therapy, including interventional chemoembolization, ablation, radiotherapy, chemotherapy, tumor palliative resection and molecular targeted therapy;
* Used any other study drugs within 5 weeks before enrollment;
* Central nervous system diseases, mental diseases, unstable angina pectoris, congestive heart failure, severe arrhythmia and other serious diseases that cannot be controlled;
* Uncontrolled infection, bleeding, pancreatic leakage, bile leakage, or other postoperative complications during baseline examination;Acute and chronic metabolic acidosis (including ketoacidosis and lactic acidosis) has not been corrected.
* A history of allergy to study drugs or similar structured drugs;
* Pregnant or lactating women;
* Any conditions, including serious medical risk factors, medical conditions, and laboratory abnormalities, that may impair patient safety or the integrity of research data;
* Intestinal obstruction, extensive adhesion in the peritoneal cavity, abdominal inflammation, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-02-23 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Ascites control | 4 weeks
  The change of abdominal volume of subjects from enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Sahnghai, China

IPD SHARING:
Plan to Share IPD: No